CLINICAL TRIAL: NCT02451527
Title: An Open-label，Single-arm，Sequential，Single-center Clinical Trial of the Pharmacokinetic Study of the Combination of Digoxin and Polythylene Glycol Loxenatide Injection (PEX168) in Healthy Adult Subjects
Brief Title: The Pharmacokinetic Study of the Combination of Digoxin and Polythylene Glycol Loxenatide Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013L02060
Record Dates: First submitted 2015-05-12; First posted 2015-05-22 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
MeSH Terms: interventions — Digoxin; polyethylene glycol loxenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Digoxin and PEX168 (Experimental): A single dose of 0.5mg digoxin administered on Day 1 followed by 5 weekly subcutaneous injections of a single dose of 200ug PEX168, followed by a further single dose of 0.5mg digoxin on Day 38.
  Interventions: Drug: Digoxin; Drug: PEX168

INTERVENTIONS:
Drug: Digoxin — Digoxin 0.5mg tablet by mouth on Day 1 and Day 38
  Other Names: Digoxine; Digoxinum; Lanoxin; Vanoxin
Drug: PEX168 — PEX168 in subcutaneous injection on Day8，15，22，29 and Day 36
  Other Names: Polythylene Glycol Loxenatide Injection

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic study of the combination of digoxin and polythylene glycol loxenatide injection (PEX168) in healthy adults，and to provide scientific basis for clinical combination of PEX168 and drugs.This study is also to evaluate the safety and tolerability of mono-digoxin or digoxin plus PEX168.

DETAILED DESCRIPTION:
This will be an open-label, single-arm, sequential, single-center clinical trial. 16 healthy males will be admitted to the clinical facility on Day -1, the day prior to the start of dosing. The subjects will be observed in clinic twice: Day -1 to 8 and Day 37 to 44. Subjects will receive a single dose of digoxin on Day 1 followed by 5 weekly subcutaneously injected doses of PEX168 and a second single dose of digoxin on Day 38. To determine the pharmacokinetic parameters of digoxin after drug administration alone and after multiple doses of PEX168, blood and urine samples will be collected after each dose of digoxin and tested by the laboratory.The subjects will be discharged on Day 8 and Day 44. Approximately 28 days after the last discharge, the subjects will be called for a post study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males aged from 18 to 45 years
2. Have a body weight over 50kg, have a body mass index (BMI) 19-25 kg/m^2 (both inclusive)
3. Alanine aminotransferase<50 U/L, aspartate aminotransferase<50 U/L, alkaline phosphatase and total bilirubin <1.5x the upper limit of normal
4. According to Cockcroft-Gault, estimated Clcr≥90ml/min
5. Able to comprehend and willing to sign the informed consent form

Exclusion Criteria:

1. Hepatitis B surface antigen(+)， Hepatitis C virus antibody(+)，AIDS antibody（+）
2. History of syncope, palpitations, bradycardia and tachycardia (for example any degree of atrioventricular block, left bundle branch block, right bundle branch block), or have an abnormal result of overall physical examination (vital signs, physical examination), routine laboratory assessment (hematology, biochemistry and urinalysis), 12-lead ECG and abdominal sonography (liver, gallbladder, pancreas, spleen, kidney)
3. Have had an alcohol and substance abuse within 6 months of screening
4. History of smoking within 3 months of screening
5. BP>140/90 millimetres of mercury, or heart rate >100 bpm
6. QT interval >450ms
7. History of drug-induced allergy or of hypersensitivity for digoxin and PEX168
8. History of serious heart disease or lung disease
9. Fasting triglyceride>1.5x the upper limit of normal
10. Subjects with liver disease or have history of liver disease or abnormal liver and gallbladder conditions
11. Donation of blood in excess of 400 mL within the 3 months of screening; or donation of blood within 1 month of screening; or received blood transfusions within 1 month of screening.
12. Hypothyroidism
13. Surgery of gastrointestinal tract
14. History of pancreatitis
15. History of cholecystitis or other gallbladder disease
16. History of inflammatory bowel disease or irritable bowel syndrome
17. History of MEN type 2 syndrome
18. History of medullary thyroid carcinoma
19. A family history of MEN type 2 syndrome and medullary thyroid carcinoma
20. Have participated in clinical trials with drug or medical devices involved within 3 months of screening
21. Have received any drug that may affect the study drugs within 2 weeks of screening, including prescribed drugs, over-counted drugs, Chinese traditional medicine or multivitamins
22. History of grapefruit juice, cranberry, mango, foods and drinks of xanthine or caffeine, strenuous exercise, or any other factor affect the absorption, distribution, metabolism and excretion of the study drug within 2 days of screening
23. Have received any glucagon-like peptide-1 mimetic compound(e.g., exenatide)
24. Have been disagreed to use a reliable method of birth control during the study and for 6 months following the last dose of study drug
25. History of any other condition, which in the opinion of the investigator, may prevent the subject from following and completing the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Composite of pharmacokinetic (PK) parameters of digoxin with and without PEX168 in plasma and urine (cmax, t 1/2) | Day 1 through Day 44
  Maximum observed concentration in plasma(cmax); apparent terminal elimination half-life in plasma(t1/2).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Day 1 through Day 44

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China